CLINICAL TRIAL: NCT01334762
Title: Letrozole and CC Alone in an IUI Program in Women With Surgically Treated Minimal to Mild Endometriosis
Brief Title: Efficacy of Letrozole and CC Alone in an IUI Program in Cases With Surgically Treated Minimal to Mild Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Dr. Hatem Abu Hashim, Associate Prof. of OB/GYN, Mansoura Faculty of Medicine, Mansoura University.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-157x; FMH-92-B
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Endometriosis
Keywords: minimal to mild endometriosis; letrozole; clomiphene citrate; IUI
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole/IUI (Experimental): Patients received 5 mg letrozole daily for 5 days. A single insemination was performed 32-36 hours after hCG (10,000 IU, IM). Patients underwent up to four cycles of treatment.
  Interventions: Drug: Letrozole/IUI
- CC/IUI (Active Comparator): Patients received 100 mg CC daily for 5 days. A single insemination was performed 32-36 hours after hCG (10,000 IU, IM). Patients underwent up to four cycles of treatment.
  Interventions: Drug: CC/IUI

INTERVENTIONS:
Drug: Letrozole/IUI — Patients received 5 mg letrozole daily for 5 days. A single insemination was performed 32-36 hours after hCG (10,000 IU, IM). Patients underwent up to four cycles of treatment.
  Arms: Letrozole/IUI
Drug: CC/IUI — Patients received 100 mg lCC daily for 5 days. A single insemination was performed 32-36 hours after hCG (10,000 IU, IM). Patients underwent up to four cycles of treatment.
  Arms: CC/IUI

SUMMARY:
To evaluate pregnancy rates with letrozole and CC alone in an IUI program for women with recently surgically treated minimal to mild endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with minimal-mild endometriosis recently treated by laparoscopy with a waiting period of 6 to 12 months following the procedure
* No other infertility factors.
* Normal serum basal hormone levels as well as documented ovulation

Exclusion Criteria:

* Moderate or severe endometriosis
* Dense adnexal and/or ovarian adhesions due to pelvic inflammatory disease or previous pelvic surgery
* Age more than 36 years, BMI more than 30 kg/m2
* women with a previous pregnancy

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate per cycle | 6-7 weeks gestation

SECONDARY OUTCOMES:
Miscarriage rate. | Up to 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD MRCOG, Principal Investigator — Mansoura University Hospital; Mohamed El Rakhawy, MD, Study Chair — Mansoura University Hospital; Ibrahim Abd Elaal, Study Director — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals,OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Dmowski WP, Pry M, Ding J, Rana N. Cycle-specific and cumulative fecundity in patients with endometriosis who are undergoing controlled ovarian hyperstimulation-intrauterine insemination or in vitro fertilization-embryo transfer. Fertil Steril. 2002 Oct;78(4):750-6. doi: 10.1016/s0015-0282(02)03343-5. PMID 12372451
- [Background] Werbrouck E, Spiessens C, Meuleman C, D'Hooghe T. No difference in cycle pregnancy rate and in cumulative live-birth rate between women with surgically treated minimal to mild endometriosis and women with unexplained infertility after controlled ovarian hyperstimulation and intrauterine insemination. Fertil Steril. 2006 Sep;86(3):566-71. doi: 10.1016/j.fertnstert.2006.01.044. PMID 16952506
- [Derived] Abu Hashim H, El Rakhawy M, Abd Elaal I. Randomized comparison of superovulation with letrozole vs. clomiphene citrate in an IUI program for women with recently surgically treated minimal to mild endometriosis. Acta Obstet Gynecol Scand. 2012 Mar;91(3):338-45. doi: 10.1111/j.1600-0412.2011.01346.x. Epub 2012 Jan 26. PMID 22181973